CLINICAL TRIAL: NCT03133221
Title: 1630GCC: A Pilot Study of Zydelig in Patients With B-cell Malignancies as Post-Autologous Transplant Remission Maintenance
Brief Title: 1630GCC: Zydelig Maintenance in B-Cell Non-Hodgkin's Lymphoma After Autologous Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Gilead Sciences (Industry); University of Miami Sylvester Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Jean A Yared, MD, Associate Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00072715; 1630GCC
Record Dates: First submitted 2017-04-13; First posted 2017-04-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Non Hodgkin Lymphoma; Follicular Lymphoma; Indolent Lymphoma; B-cell Lymphoma; Transformed Lymphoma; Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia; Small Lymphocytic Lymphoma; Lymphoplasmacytic Lymphoma
Keywords: NHL; indolent NHL; Zydelig; Idelalisib; B-cell NHL; Non-Hodgkin Lymphoma; Maintenance; Transformed B-cell Non-Hodgkin's lymphoma; Autologous Stem Cell Transplantation
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Zydelig 150 mg BID (Experimental): Zydelig given orally at 150 mg twice daily continuously on 28-day cycles starting 30 to 120 days after autologous stem cell transplantation for patients with indolent or transformed indolent B-cell NHL, for up to 1 year maintenance duration. Dose withhold/modification is allowed according to tolerability/toxicity.
  Interventions: Drug: Zydelig

INTERVENTIONS:
Drug: Zydelig — Zydelig given at 150mg continuously in 28-day cycles
  Other Names: Idelalisib

SUMMARY:
This is a pilot study to learn how safe and how effective the study drug Zydelig works, after autologous stem cell transplant as a maintenance therapy in patients with indolent or transformed indolent B-cell non-Hodgkins lymphoma (iNHL or tiNHL).

DETAILED DESCRIPTION:
This pilot study is focused on maintenance Zydelig for patients with indolent or transformed indolent B-cell non-Hodgkins lymphoma (iNHL or tiNHL) after autologous stem cell transplantation. Oral Zydelig at 150 mg (or adjusted dose) twice daily continuously on 28-day cycles. Patients will continue on Zydelig up to one year or to progression/relapse/death or unacceptable toxicity, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented (by HPI or pathology report) iNHL as defined by follicular lymphoma (FL), marginal zone lymphoma (MZL), lymphoplasmacytic lymphoma/Waldenstrom disease (LPL/WM) and small lymphocytic lymphoma (SLL) or tiNHL as defined by large B cell transformation of any of the above entities including chronic lymphocytic leukemia (CLL)
2. Patients must be eligible to undergo high dose chemotherapy (HDT) followed by ASCT as a form of remission consolidation
3. Patients without evidence of documented disease progression clinically or radiographically after ASCT (stable disease (SD), partial remission (PR) or complete remission (CR)) who have had count recovery (ANC > 500, non-transfused platelet count > 20,000) and are at least 30 days post ASCT but no more than 120 days post ASCT
4. Patients may have received any prior therapy deemed necessary for them to be eligible to HDT/ASCT except for patients whom have progressed while on Zydelig. Patients who have responded to Zydelig previously are eligible for enrollment on the protocol.
5. Age >18
6. ECOG performance status <4
7. Life expectancy of greater than four months.
8. Patients must have normal organ function as defined below (after the HDT/ASCT):

   * total bilirubin less than 2x institutional upper limit of normal
   * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
   * Creatinine < 1.5x institutional upper limit of normal OR creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels > 1.5x upper limit of normal.
9. Because the effects of Zydelig on the developing human fetus are unknown, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Participants must agree to use contraception for at least 30 days after the last dose of Zydelig. Women of childbearing potential is defined as women who continues to have menstrual periods, have not had a tubal ligation, or the removal of fallopian tubes, ovaries or uterus.
10. Ability to understand English and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 2 weeks of first dose of Zydelig.
2. Patients receiving any other investigational agents within 30 days of receiving Zydelig
3. Patients who were previously exposed to Zydelig and experienced progression of disease.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Zydelig.
5. Patients with active and/or untreated CNS lymphoma will not be eligible.
6. Patients with inflammatory bowel disease.
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection (defined as requiring systemic antibiotic treatment and fever within 48 hours of screening), symptomatic congestive heart failure (patients with NYHA score of III and above are excluded), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Women who are pregnant or nursing or plan to become pregnant or nurse during the course of the study.
9. Positive HIV status.
10. Patients with lack of count recovery as defined in Protocol 3.1.1.1.1.
11. Patients who are unable to swallow pills.
12. Patients with moderate to severe lung disease including:

    * Patients requiring O2 supplementation
    * Patients unable to walk 50 feet without stopping to rest
    * Moderate to severe obstructive or restrictive disease of the lung
13. Patients taking strong CYP3A4 inhibitors or inducers with Risk X (Avoid Combination) according to Lexicomp. Please see appendix C of the protocol for more information.
14. Patients with active hepatic disease, liver cirrhosis, or known HBV/HCV infection.
15. Patients with de novo diffuse large B-cell lymphoma.
16. Patients with h/o PCP pneumonia or CMV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Yared, MD, Principal Investigator — University of Maryland Greenebaum Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Zydelig 150 mg BID
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oral Zydelig 150 mg BID
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 60.82 [44.98 to 72.49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Discontinuation Rate Due to Zydelig-related Adverse Events at 1 Year
Description: The proportion of patients who discontinued the study due to Zydelig-related adverse events.
Time Frame: 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Zydelig 150 mg BID
Number analyzed (Participants) | 17
Participants | 5

2. Secondary Outcome: Progression-free Survival at 1 and 2 Years After Autologous Stem Cell Transplantation.
Description: 1- and 2-year Progression-free survival; Progression-free survival is defined as time from the date of autologous stem cell transplantation to progression, relapse and death, whichever comes first.
Time Frame: 1- and 2-year Progression-free survival
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Zydelig 150 mg BID
Number analyzed (Participants) | 17
Participants
  Progression-free survival | 13
  1 year post transplant relapse | 1
  2 year post transplant relapse | 3

ADVERSE EVENTS:
Time Frame: 2 years post Autologous Stem Cell Transplantation (HDT/ASCT)
Arm/Group | Oral Zydelig 150 mg BID
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 9/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Zydelig 150 mg BID (N=17)
Diarrhea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Zydelig 150 mg BID (N=17)
Abdominal Pain (General disorders) | 2
Acute bilateral maxillary sinusitis (Infections and infestations) | 1
Alkaline Phosphatase Increased (Blood and lymphatic system disorders) | 1
ALT Decreased (Blood and lymphatic system disorders) | 1
ALT increase (Blood and lymphatic system disorders) | 4
Anorexia (General disorders) | 1
Arthralgia (General disorders) | 2
AST Decreased (Blood and lymphatic system disorders) | 1
AST Increase (Blood and lymphatic system disorders) | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (General disorders) | 1
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1
Bruising (General disorders) | 1
Chills (General disorders) | 2
Conjunctival erythema (Eye disorders) | 1
Conjunctival irritation (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (General disorders) | 5
Creatinine decreased (Blood and lymphatic system disorders) | 1
Creatinine increased (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dry eyes (Ear and labyrinth disorders) | 1
Dysgeusia (General disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Dyspnea (General disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Headache (General disorders) | 2
Hemoglobin Decreased (Blood and lymphatic system disorders) | 6
Herpatoxicity (Gastrointestinal disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 7
Hyperuricemia (Blood and lymphatic system disorders) | 2
Hypocalcemia (Blood and lymphatic system disorders) | 1
Hypoglycemia (Blood and lymphatic system disorders) | 1
Hypokalemia (Blood and lymphatic system disorders) | 1
Hypomagnesemia (Blood and lymphatic system disorders) | 1
IgG deficiency (Blood and lymphatic system disorders) | 1
Insomnia (General disorders) | 5
Irritability (General disorders) | 1
Lacerations (feet) (Skin and subcutaneous tissue disorders) | 1
LDH decrease (Blood and lymphatic system disorders) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1
Mouth sore (General disorders) | 2
Nail discoloration (General disorders) | 2
Nausea (General disorders) | 4
Neutrophils decreased (Blood and lymphatic system disorders) | 5
Night sweats (General disorders) | 1
Pain in extremities (General disorders) | 1
Peripheral Edema (Skin and subcutaneous tissue disorders) | 2
Peripheral neuropathy (Skin and subcutaneous tissue disorders) | 1
Platelets decreased (Blood and lymphatic system disorders) | 7
Pleuritic chest pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Proctitis (Gastrointestinal disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 9
Renal insufficiency (Renal and urinary disorders) | 1
Restless leg syndrome (General disorders) | 1
Scalp lesion (Skin and subcutaneous tissue disorders) | 1
Sinusitis (General disorders) | 1
Sore throat (General disorders) | 1
Transaminitis (Blood and lymphatic system disorders) | 4
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5
Urinary incontinence (Endocrine disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
WBC Decreased (Blood and lymphatic system disorders) | 6
Weight loss (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT03133221/Prot_SAP_000.pdf